CLINICAL TRIAL: NCT04246840
Title: Study Through Imaging of Mediastinal and Abdominopelvic Secondary Lymphoid Organs (Lymph Nodes) in Patients With Severe Combined Immunodeficiencies (SCID) Who Have Recieved Bone Narrow Allograft
Brief Title: Study Through Imaging of Visceral Lymphoid Organs in Patients With SCID Who Have Recieved Bone Marrow Allograft
Acronym: LymphImaging
Status: Completed | Type: Observational
Sponsor: Association Pour l'Aide a la Recherche en Immunologie Pediatrique (Other)
Responsible Party: Sponsor
Other Study IDs: AARIP-01
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Severe Combined Immunodeficiency
MeSH Terms: conditions — Severe Combined Immunodeficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: 15 adult patients who underwent allogenic hematopoietic stem cell transplantation (HSCT) for severe combined immunodeficieny 15 to 45 years ago
- Control group: 15 age-matched healthy individuals

SUMMARY:
To investigate the presence of seconday of lymphoid organs in patients who underwent allogenic hematopoietic stem cell transplantation 15 to 45 years ago.

The goal aims to assess the development of seconday lymphoid organs given the fact that the absence of myeloablation these patients present a split chimerism between T lymphocytes and the other leucocytes. Thus, they may not be able to generate seconday lymphoid organs. Practically, whole body MRI is being used to visualise and quantify both mediastinal and intraabdominal lymph nodes. Delta will be compared with those obtained in healthy age-matched individuals. It is scheduled to include 15 patients and 15 controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SCID transplanted 15-45 years ago

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with SCID transplanted 15-45 years ago and healthy conrtrols
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Size of mediastinal and intraabdominal lymph nodes | 1 year
  analysis by MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Necker, Paris, France

REFERENCES:
- [Derived] Berteloot L, Molina TJ, Bruneau J, Picard C, Barlogis V, Secq V, Abdo C, Boddaert N, Griscelli C, Neven B, Fischer A. Alternative pathways for the development of lymphoid structures in humans. Proc Natl Acad Sci U S A. 2021 Jul 20;118(29):e2108082118. doi: 10.1073/pnas.2108082118. PMID 34261794